CLINICAL TRIAL: NCT04750148
Title: Comparison of the 2MWT, the 10MeWT and the 6MWT in Individuals With Cancer, a Validation Observational Study.
Brief Title: Validation of the Two-minute Walk Test and the Ten-meter Walk Test in Individuals With Cancer
Acronym: 2MWTOnco
Status: Completed | Type: Observational
Sponsor: Aline Reinmann (Other)
Responsible Party: Sponsor-Investigator, Aline Reinmann, Principal Investigator, School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Other Study IDs: 2020-00126
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Cancer
Keywords: 6-minute walking test; 2-minute walking test; 10-meter walk test
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer: Individuals with an oncology disease will be included in the study.
  Interventions: Diagnostic Test: 6-minute walking test; Diagnostic Test: 2-minute walking test; Diagnostic Test: 10-meter walk test; Diagnostic Test: One leg stance test

INTERVENTIONS:
Diagnostic Test: 6-minute walking test — The subject walks as far as possible for 6 minutes along a 30m long corridor.
Diagnostic Test: 2-minute walking test — The subject walks as far as possible for 2 minutes along a 30m long corridor.
Diagnostic Test: 10-meter walk test — The natural and fast walking speeds of the subject are measured over 10m. This speed is measured by the examiner as well as by the subject (self-tested version).
Diagnostic Test: One leg stance test — The time held in unipodal equilibrium is measured by the examiner.

SUMMARY:
The aim of this study is to assess the feasibility and the validity of the 2-minute walk test (2MWT) and the 10-meter walk test (10MeWT) compared to the 6-minute walk test (6MWT) for subjects with onco-hematological disease.

DETAILED DESCRIPTION:
Cancer and its treatments have an impact on the body as a whole. The analysis of the subject's physical capacity is essential to know the basic level of the subject pre-treatment, to evaluate progress following rehabilitation, to set goals to prevent decline in physical capacity or to evaluate changes in physical capacity at different stages of survival. The 6-minute walk test (6MWT) is frequently used in the clinic to assess the physical capacity of the subject in oncology. A variant of the 6MWT exists and has been little studied in an oncological context: the 2-minute walk test (2MWT). The 2MWT is performed in the same way as the 6MWT: the same instructions and the same test procedure. It offers the advantage of being less tiring for the test subjects and saves clinicians time. The 2MWT has been validated in the past for people with COPD or after cardiac surgery. To our knowledge, it has not been validated for cancer patients.

The 10-meter walk test (10MeWT) is frequently used in practice to assess patients' functional capacity. It would be another way to assess the walking ability with a short test.

However, the relationship between the 2MWT, 6MWT and 10MeWT in an oncological context remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* Have an onco-hematologic disease
* Have medical authorization from the patient's oncologist authorizing gait tests
* Participate in the HUG rehabilitation program
* Be able to give consent by signature
* To be of legal age
* Do not present pain when walking more than 2/10
* Be able to walk with or without technical aids for a period of 6 minutes (as per patient's statement)

Exclusion Criteria:

* Suffer from heart problems
* Bone metastases at risk of fracture
* Osteoporosis at high risk of fracture
* Unbalanced Hypertension (hypertension)
* Not being able to carry out the walk tests in their entirety
* Not being able to perform the gait tests for reasons related to the side effects of the treatments (anemia, undernutrition, vomiting, severe fatigue, risk of thrombocytopenia, pain).
* Not being able to carry out the walking test because of a lack of understanding of the instructions or because of psychological problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 50 adults consulting at the University Hospitals for their oncological disease.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: feasibility of the 2MWT and the 10MeWT | through study completion, an average of 1 year
  The feasibility of the different tests will be assessed in an oncological setting.
Primary endpoint: criterion validity with the 6MWT | through study completion, an average of 1 year
  Criterion validity will be assessed by calculating the strength of the correlation between the 2MWT/10MeWT and the 6MWT.

SECONDARY OUTCOMES:
Secondary endpoint: convergent construct validity | through study completion, an average of 1 year
  Convergent construct validity will be evaluated by calculating the strength of the correlation between the 2MWT and the 10m walk test at comfortable/fast speed
Secondary endpoint: criterion validity between 10m walk test and 10m walk test self-tested | through study completion, an average of 1 year
  Criterion validity will be assessed by calculating the strength of the correlation between the 10m walk test self-tested and the 10m walk test timed by the examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Reinmann, Principal Investigator — School of Health Sciences Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes will be made available.
Time Frame: Data will be available within 6 months of study completion

REFERENCES:
- [Background] Bohannon RW, Bubela D, Magasi S, McCreath H, Wang YC, Reuben D, Rymer WZ, Gershon R. Comparison of walking performance over the first 2 minutes and the full 6 minutes of the Six-Minute Walk Test. BMC Res Notes. 2014 Apr 25;7:269. doi: 10.1186/1756-0500-7-269. PMID 24767634
- [Background] Butland RJ, Pang J, Gross ER, Woodcock AA, Geddes DM. Two-, six-, and 12-minute walking tests in respiratory disease. Br Med J (Clin Res Ed). 1982 May 29;284(6329):1607-8. doi: 10.1136/bmj.284.6329.1607. No abstract available. PMID 6805625
- [Background] Chan WLS, Pin TW. Reliability, validity and minimal detectable change of 2-minute walk test, 6-minute walk test and 10-meter walk test in frail older adults with dementia. Exp Gerontol. 2019 Jan;115:9-18. doi: 10.1016/j.exger.2018.11.001. Epub 2018 Nov 10. PMID 30423359
- [Background] Eden MM, Tompkins J, Verheijde JL. Reliability and a correlational analysis of the 6MWT, ten-meter walk test, thirty second sit to stand, and the linear analog scale of function in patients with head and neck cancer. Physiother Theory Pract. 2018 Mar;34(3):202-211. doi: 10.1080/09593985.2017.1390803. Epub 2017 Oct 25. PMID 29068767
- [Background] Gijbels D, Eijnde BO, Feys P. Comparison of the 2- and 6-minute walk test in multiple sclerosis. Mult Scler. 2011 Oct;17(10):1269-72. doi: 10.1177/1352458511408475. Epub 2011 Jun 3. PMID 21642370
- [Background] Kosak M, Smith T. Comparison of the 2-, 6-, and 12-minute walk tests in patients with stroke. J Rehabil Res Dev. 2005 Jan-Feb;42(1):103-7. doi: 10.1682/jrrd.2003.11.0171. PMID 15742254
- [Background] Leung AS, Chan KK, Sykes K, Chan KS. Reliability, validity, and responsiveness of a 2-min walk test to assess exercise capacity of COPD patients. Chest. 2006 Jul;130(1):119-25. doi: 10.1378/chest.130.1.119. PMID 16840391
- [Background] Reid L, Thomson P, Besemann M, Dudek N. Going places: Does the two-minute walk test predict the six-minute walk test in lower extremity amputees? J Rehabil Med. 2015 Mar;47(3):256-61. doi: 10.2340/16501977-1916. PMID 25588644
- [Background] Scalzitti DA, Harwood KJ, Maring JR, Leach SJ, Ruckert EA, Costello E. Validation of the 2-Minute Walk Test with the 6-Minute Walk Test and Other Functional Measures in Persons with Multiple Sclerosis. Int J MS Care. 2018 Jul-Aug;20(4):158-163. doi: 10.7224/1537-2073.2017-046. PMID 30150899
- [Background] Schmidt K, Vogt L, Thiel C, Jager E, Banzer W. Validity of the six-minute walk test in cancer patients. Int J Sports Med. 2013 Jul;34(7):631-6. doi: 10.1055/s-0032-1323746. Epub 2013 Feb 26. PMID 23444095